CLINICAL TRIAL: NCT05786937
Title: Therapeutic Vaccine Based on aDC1 Dendritic Cells for the Control of Viremia After Antiretroviral Therapy Interruption in HIV Infected Individuals
Brief Title: Therapeutic Vaccine Based on aDC1 Dendritic Cells for the Control of Viremia After ATI in HIV Infected Individuals
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Alberto José da Silva Duarte, Professor Doctor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INHC031
Record Dates: First submitted 2023-03-14; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: HIV Vaccine
Keywords: HIV; Immunotherapy; Polarizing dendritic cells
MeSH Terms: interventions — Heart Rate

STUDY DESIGN:
Intervention Model Description: Phase I, double-blind, randomized study with three parallel groups as follows: : G1) placebo; G2) aDC1immunization; G3) aDC1 immunization with analytical treatment interruption of ART.
Who Masked: Participant, Care Provider
Masking Description: To avoid bias in evaluating the results, the research volunteer and the team that will perform the application of the vaccine product will be blind in the present study. The team responsible for coordinating the project will not be blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): The participants will receive a placebo, which is the excipient solution of aDC1 cell suspension consisting of a commercial ringer´s lactate solution.
  Interventions: Other: Commercial ringer´s lactate solution
- aDC1immunization (Active Comparator): The participants will be immunized with aDC1 unpulsed with HIV peptides.
  Interventions: Biological: Alpha-type-1 Polarizing Dendritic Cells (aDC1) unpulsed with HIV peptides
- aDC1 immunization with analytical treatment interruption of ART (Experimental): The participants will be immunized with aDC1 pulsed with HIV peptides.
  Interventions: Biological: Alpha-type-1 Polarizing Dendritic Cells (aDC1) pulsed with HIV peptides

INTERVENTIONS:
Biological: Alpha-type-1 Polarizing Dendritic Cells (aDC1) unpulsed with HIV peptides — Alpha-type-1 Polarizing Dendritic Cells (aDC1) unpulsed with HIV peptides
  Arms: aDC1immunization
Biological: Alpha-type-1 Polarizing Dendritic Cells (aDC1) pulsed with HIV peptides — Alpha-type-1 Polarizing Dendritic Cells (aDC1) pulsed with HIV peptides
  Arms: aDC1 immunization with analytical treatment interruption of ART
Other: Commercial ringer´s lactate solution — Placebo
  Arms: Placebo

SUMMARY:
The goal of this interventional study is to validate the strategy of adjuvant therapy with dendritic cells in HIV infection in chronically infected individuals. The main questions it aims to answer are related to the safety and tolerance of the intervention and the virological and immunological impact of immunotherapy with aDC1 in HIV-infected individuals. The study will include 30 diagnosed HIV-infected patients, using antiretroviral therapy, who will be immunized with aDC1 or placebo according to the arms of this study: G1) placebo; G2) aDC1immunization; G3) aDC1 immunization with analytical treatment interruption of ART.

DETAILED DESCRIPTION:
Dendritic cell based immunotherapy is a potential tool to stimulate a specific immune response, as a complementary treatment for HIV-infected individuals using ART. Polarizing DCs are capable to produce high levels of IL-12p70 and induce a strong cytotoxic response that is very useful in viral infections. In this context, we propose to study aDC1 pulsed with relevant HIV peptides for treatment of HIV infected individuals.

The study will include 30 diagnosed HIV-infected patients, using antiretroviral therapy, who will be immunized with aDC1 or placebo according to the arms of this study: G1) placebo; G2) aDC1immunization; G3) aDC1 immunization with analytical treatment interruption of ART. Autologous PBMCs will be collected for baseline parameters and vaccine will be inoculated in 3 doses (with 4 week interval). Three weeks after 3th vaccine inoculation, patients will be followed for 6 months and blood and biopsis samples will be collected for different parameters measurement as immune activation, immunogenicity, humoral response, mucosal cellular immunity and virologic profile and viral reservoir analysis.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection confirmed according to the criteria of the Department of Chronic Diseases and Sexually Transmitted Infections of the Brazilian Health Ministry;
* Absence of the use of antineoplastic or corticosteroid therapies for a minimum period of six months prior to study entry;
* Absence of comorbidities considered uncontrolled by researchers;
* Viral load ≤ 40 copies/mL, stable (i.e., no > 0.5 log) in the six months prior to the start of the study;
* Blood count of CD4 T lymphocytes ≥ 500 cells/μL, stable (i.e., >25%) in the six months prior to the start of the study;
* Informed consent

Exclusion Criteria:

* Individuals without adequate venous access to the blood collection and apheresis procedure;
* Use of drugs or alcohol in a way that interferes with patients' ability to follow the study requirements;
* Pregnancy, breastfeeding or interest in becoming pregnant during the study period;
* Presence of any other condition that, in the evaluation of researchers is able to promote alteration of the immune system, as well as any disorders that could affect understanding in the process of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events related to the study product | Six months
  Number of participants with adverse events related to the study product
Plasma viral load setpoint after the intervention | Six months
  Number of participants with changes in the plasma viral load setpoint after the intervention
Setpoint of CD4+ T lymphocyte count after the intervention | Six months
  Number of participants with changes in the setpoint of CD4+ T lymphocyte count after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alberto José DS Duarte, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No